CLINICAL TRIAL: NCT03834311
Title: The Effectiveness of Upper Extremity Isokinetic Strengthening in Post-stroke Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ilke Coskun Benlidayi, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CukurovaPMR
Record Dates: First submitted 2019-01-06; First posted 2019-02-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stroke Rehabilitation; Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- isokinetic (Experimental)
  Interventions: Device: isokinetic strengthening
- exercise band (Active Comparator)
  Interventions: Other: exercise band strengthening

INTERVENTIONS:
Device: isokinetic strengthening — isokinetic upper extremity (forearm) strengthening for 4 weeks 3d/w
  Arms: isokinetic
Other: exercise band strengthening — upper extremity (forearm) strengthening with exercise band 4 weeks 3d/w
  Arms: exercise band

SUMMARY:
This randomised controlled study will investigate the effectiveness of isokinetic strengthening on the upper extremity functionality and strength in post-stroke hemiplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* Active motion in upper extremity
* Brunnstrom's Scale above 3

Exclusion Criteria:

* Unstable medical conditions
* Cognitive problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
upper extremity strength | 0, 4, 8 weeks (change from baseline upper extremity strength at 4 weeks and at 8 weeks will be assessed)
  Muscles: forearm flexors and extensors Measurement tool: MicroFET3 (Hoggan Health Industries Inc. West Jordan, UT, USA)
pik torque | 0, 4, 8 weeks (change from baseline pik torque at 4 weeks and at 8 weeks will be assessed)
  Muscles: wrist flexors and extensors Measurement Tool: CSMI Humac Norm Cybex isokinetic dinamometer (HUMAC® /2009 Version: 10.000.0065, Computer Sports Medicine Inc., USA)

SECONDARY OUTCOMES:
hand grip strength | 0, 4, 8 weeks
  Measurement tool: Jamar Hydraulic Hand Dynamometer (Patterson Medical, Warrenville, IL, USA)
Fugl-Meyer Assessment scale for upper extremity | 0, 4, 8 weeks
  Scale range: 0-66; higher values represent a better outcome; subscales are combined by summing to compute a total score
Disabilities of the arm, shoulder and hand questionnaire (Part 1) | 0, 4, 8 weeks
  Scale range: 0-100; higher scores represent more disabilities of the upper limb; Total score (sum of the scores for 30 questions) is put in a formula to compute the DASH disability score
Stroke Impact Scale version 3.0 | 0, 4, 8 weeks
  Includes 8 domains and an extra assessment for stroke recovery; scores range 0-100 for each domain; higher scores represent better outcome; a formula is used for scoring each domain.

CONTACTS AND LOCATIONS:
Locations (1):
- İlke COŞKUN BENLİDAYI, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kerimov K, Coskun Benlidayi I, Ozdemir C, Gunasti O. The Effects of Upper Extremity Isokinetic Strengthening in Post-Stroke Hemiplegia: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2021 Jun;30(6):105729. doi: 10.1016/j.jstrokecerebrovasdis.2021.105729. Epub 2021 Mar 23. PMID 33765633